CLINICAL TRIAL: NCT00103545
Title: A Phase I/II Trial of ACA 125 in Patients With Recurrent Epithelial Ovarian, Fallopian Tube or Peritoneal Cancer
Brief Title: Use of ACA 125 in Patients With Ovarian Cancer: Safety and Immune Response
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGO-OVAR 2.8
Record Dates: First submitted 2005-02-10; First posted 2005-02-11 (Estimated); Last update posted 2006-10-02 (Estimated); Status verified 2006-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: Ovarian Cancer; ACA 125; 6 or 9 vaccinations; immune response; Fallopian tube cancer; Peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — abagovomab

INTERVENTIONS:
Biological: ACA 125

SUMMARY:
The purpose of this study is to use an immunologic approach following the treatment for recurrent disease in patients with ovarian, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
Patients with epithelial ovarian, fallopian tube or peritoneal cancer who receive surgical cytoreduction and platinum/taxane containing chemotherapy have a significant chance of entering complete clinical remission but about 70% will eventually relapse. Many patients respond to additional cytotoxic treatment with partial or complete responses, yet approximately 100% of these patients will ultimately progress. Novel consolidation strategies following treatment for recurrent disease are needed and an immunologic approach is an attractive option.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epithelial carcinoma arising in the ovary, fallopian tube or peritoneum, stages I-IV. These patients must have received initial surgery and chemotherapy with at least one platinum based chemotherapy regimen.
* Patients must have relapsed and now have completed chemotherapy for recurrent disease within the last 6 weeks.
* Eligible patients may have asymptomatic residual measurable disease on CT scan, and/or may have an elevated CA-125, or may be in complete clinical remission.
* Patients must have adequate hematologic, renal and hepatic functions.

Exclusion Criteria:

* Patients with any other active malignancy concomitantly
* Patients within 3 weeks of prior cytotoxic or investigational chemotherapy
* Patients within 4 weeks of prior radiotherapy
* Patients within 6 weeks of prior immunotherapy
* Patients who have received any prior anti-cancer vaccine

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Start 2003-07; Study Completion 2004-08

PRIMARY OUTCOMES:
Safety, feasibility and tolerability
The primary endpoint is drop-out due to toxicity as the overall measure of feasibility

SECONDARY OUTCOMES:
Duration and strength of the immune response induced by ACA 125 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus Pfisterer, Prof. Dr., Principal Investigator — AGO Study Group
Locations (11):
- Germany (11):
  - Clinic for Gynecology and Gyn. Oncology, Humboldt University, Berlin
  - University Clinic Carl Gustav Carus, Gynecological hospital, Dresden
  - Gynecologic Hospital, Düsseldorf
  - University Gynecologic Hospital, Essen
  - University Gynecologic Hospital, Frankfurt
  - Gynecologic Clinic of the Ernst-Moritz-Arndt-University, Greifswald
  - University Clinic Schleswig-Holstein, Campus Kiel, Clinic for gynecology and obstetrics, Kiel
  - Otto-von-Guericke University, University Gynecological Hospital, Magdeburg
  - Clinic of the Philipps University Marburg, Clinic for gynecology, gyn. endocrinology and oncology, Marburg
  - University Gynecological Hospital, Ulm
  - Clinic for Gnyecology and gyn. Oncology HSK, Wiesbaden

REFERENCES:
- [Background] Pfisterer J, du Bois A, Sehouli J, Loibl S, Reinartz S, Reuss A, Canzler U, Belau A, Jackisch C, Kimmig R, Wollschlaeger K, Heilmann V, Hilpert F. The anti-idiotypic antibody abagovomab in patients with recurrent ovarian cancer. A phase I trial of the AGO-OVAR. Ann Oncol. 2006 Oct;17(10):1568-77. doi: 10.1093/annonc/mdl357. PMID 17005631
- See also: Information on studies of the AGO-OVAR on Ovarian cancer — http://www.ago-ovar.de